CLINICAL TRIAL: NCT00364533
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Multiple Doses of CG5503 Immediate Release Formulation in the Treatment of Acute Pain From Total Hip Replacement Surgery Followed by a Voluntary Open-Label Extension
Brief Title: A Study to Evaluate the Effectiveness and Safety of Tapentadol(CG5503) in the Treatment of Acute Pain After Hip Replacement Surgery Compared With Oxycodone and Placebo Followed by a Voluntary Open-Label Extension For Safety
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR011221; R331333PAI3001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); KF5503/31 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Arthroplasty
Keywords: Arthralgia; Pain; Pain Assessment; Hip Replacement; Tapentadol
MeSH Terms: conditions — Arthralgia; Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 003 (Placebo Comparator): Placebo Fixed Dose Matching placebo for 3 days
  Interventions: Drug: Placebo
- 002 (Active Comparator): Oxycodone HCL IR Fixed Dose 10 mg BID for 3 days
  Interventions: Drug: Oxycodone HCL IR
- 001 (Experimental): Tapentadol IR (CG5503) Fixed Dose 50, 75, & 100 mg BID for 3 days
  Interventions: Drug: Tapentadol IR (CG5503)
- 004 (Other): Tapentadol IR (CG5503) Flexible Dose q4-6 hr Tapentadol IR 50 & 100 mg BID for 9 days
  Interventions: Drug: Tapentadol IR (CG5503)

INTERVENTIONS:
Drug: Tapentadol IR (CG5503) — Fixed Dose 50, 75, & 100 mg BID for 3 days
  Arms: 001
Drug: Placebo — Fixed Dose Matching placebo for 3 days
  Arms: 003
Drug: Oxycodone HCL IR — Fixed Dose 10 mg BID for 3 days
  Arms: 002
Drug: Tapentadol IR (CG5503) — Flexible Dose q4-6 hr Tapentadol IR 50 & 100 mg BID for 9 days
  Arms: 004

SUMMARY:
The purpose of this study is to test in patients who have had hip replacement surgery the effectiveness (level of pain control) and the safety of 3 different dose levels of CG5503 compared with placebo and with 10-mg oxycodone during the 72-hour double-blind period and to assess the safety of the drug for 9 days after patients completed the double blind period.

DETAILED DESCRIPTION:
Patients undergoing hip replacement often experience moderate to severe acute pain post-surgery. Normally such pain is controlled when patients receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, addiction, tolerance, and respiratory depression. CG5503, a newly synthesized drug also acts as a centrally acting pain reliever but has a dual mode of action. The aim of this study is to investigate the effectiveness (level of pain control) and safety (side effects) of 3 dose levels of CG5503, in an immediate release, (IR) formulation, compared with no drug (placebo) or one dose level of oxycodone (an opioid commonly used to treat post-surgical pain). This study is a randomized, double-blind (neither investigator nor patient will know which treatment was received), active- and placebo-controlled, parallel-group, multicenter study to evaluate the treatment of acute pain from hip replacement surgery. The study will include a blinded 72 hour in-patient phase immediately following hip replacement surgery, during which patients will be treated with either 50-, 75-, or 100-mg CG5503 base IR, a placebo, or 10-mg oxycodone, and pain relief will be periodically assessed. Following this phase, patients wishing to continue treatment with CG5503 IR may enter an outpatient voluntary nonrandomized, open-label extension phase for 9 days during which they will receive 50- or 100-mg CG5503 IR. Assessments of pain relief include the pain intensity numeric rating scale (PI), pain relief numeric rating scale (PAR) and patient global impression of change scale (PGIC). Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Venous blood samples will be collected for the determination of serum concentrations of CG5503 and oxycodone. The null hypothesis for the study is that efficacy results for all CG5503 IR dosage groups are equal to placebo based on the mean sum of pain intensity difference at 48 hours. The alternative study hypothesis is that at least 1 dose strength of CG5503 will be different from placebo in controlling pain at 48 hours. CG5503 base IR 50, or 75, or 100 mg, or oxycodone 10 mg, or placebo, 1 capsule taken by mouth every 4 to 6 hours during the 72 hour postsurgery phase of the study (one extra dose is allowed, if needed for pain); and CG5503, 50 mg base capsules, 1 to 2 tablets taken by mouth every 4 to 6 hours for up to 9 days during the open label portion of the study. All doses of study treatment will be taken with approximately 120 mL of water with or with food.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo standard primary (first-time) one-sided total hip replacement surgery due to degenerative joint disease (arthritis), not due to some inflammatory process, (eg. infection)
* Baseline pain intensity >= 4 on an 11-point (0 to 10) Pain Intensity rating scale, rated within 30 minutes before randomization
* Women must be postmenopausal, surgically sterile, or practicing or agree to practice an effective method of birth control throughout the study

Exclusion Criteria:

* Patients will be excluded from the study if they have a history of seizure disorder or epilepsy
* history of malignancy within the past 2 years before starting the study
* history of alcohol or drug abuse
* evidence of active infections that may spread to other areas of the body
* clinical laboratory values reflecting moderate or severe kidney insufficiency
* currently treated with anticonvulsants, monoamine oxidase inhibitors, tricyclic antidepressants, neuroleptics, or selective norepinephrine reuptake inhibitor (SNRI), (selective serotonin reuptake inhibitor [SSRI] treatments are allowed if taken for at least 30 days before the screening period of the study at an unchanged dose)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (77):
- United States (45):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Sheffield, Alabama
  - Phoenix, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Arcadia, California
  - Glendale, California
  - Laguna Hills, California
  - Sacramento, California
  - San Francisco, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Boynton Beach, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Plantation, Florida
  - Port Orange, Florida
  - Tamarac, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Topeka, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Royal Oak, Michigan
  - Albany, New York
  - Mineola, New York
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Sewickley, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Plano, Texas
  - Murray, Utah
  - Weston, Wisconsin
- Belgium (4):
  - Aalst
  - Genk
  - Ghent
  - Leuven
- Canada (9):
  - Halifax, Nova Scotia
  - Burlington, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Scarborough Village, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - London
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- Hamilton, New Zealand
- Spain (3):
  - Cadiz
  - Madrid
  - Valencia
- Sweden (4):
  - Borås
  - Hässleholm
  - Örebro
  - Uppsala
- United Kingdom (8):
  - Aberdeen
  - Birmingham
  - Edinburgh
  - Great Yarmouth
  - London
  - Middlesex
  - Sheffield
  - Wigan

REFERENCES:
- See also: A Study to Evaluate the Effectiveness and Safety of Tapentadol(CG5503) in the Treatment of Acute Pain After Hip Replacement Surgery Compared With Oxycodone and Placebo Followed by a Voluntary Open-Label Extension For Safety — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=61&filename=CR011221_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Tapentadol IR Fixed Dose 50 mg; Tapentadol IR Fixed Dose 75 mg; Tapentadol IR Fixed Dose 100 mg: Tapentadol taken by mouth every 4-6 hours for 3 days
- Oxycodone HCL IR Fixed Dose 10 mg: oxycodone 10mg taken by mouth every 4-6 hours for 3 days
- Placebo Fixed Dose: Matching placebo taken by mouth every 4-6 hours for 3 days
Period: Overall Study
Arm/Group | Tapentadol IR Fixed Dose 50 mg | Tapentadol IR Fixed Dose 75 mg | Tapentadol IR Fixed Dose 100 mg | Oxycodone HCL IR Fixed Dose 10 mg | Placebo Fixed Dose
Started | 77 | 71 | 75 | 67 | 75
Completed | 35 | 31 | 30 | 36 | 24
Not Completed | 42 | 40 | 45 | 31 | 51
Not completed — Adverse Event | 8 | 7 | 15 | 5 | 2
Not completed — Withdrawal by Subject | 4 | 8 | 6 | 6 | 6
Not completed — Lack of Efficacy | 22 | 22 | 21 | 17 | 42
Not completed — Subject discharged from hospital | 4 | 1 | 2 | 3 | 1
Not completed — Variations in drug compliance | 2 | 1 | 1 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol IR Fixed Dose 50 mg | Tapentadol IR Fixed Dose 75 mg | Tapentadol IR Fixed Dose 100 mg | Oxycodone HCL IR Fixed Dose 10 mg | Placebo Fixed Dose | Total
Number analyzed (Participants) | 77 | 71 | 75 | 67 | 75 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.20) | 62.8 (9.24) | 63.3 (10.3) | 61.3 (12.39) | 64.0 (11.23) | 62.7 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 32 | 41 | 41 | 44 | 197
  Male | 38 | 39 | 34 | 26 | 31 | 168

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference Over 48 Hours (SPID48)
Description: The SPID score incorporates the cumulative analgesic effects of tapentadol IR on pain intensity over an extended period (48 hours) allowing for an evaluation of multiple doses of drug, even when dosing frequency may vary. Scoring is derived from the Numerical Rating Scale (NRS) from 0 = No pain to 11 = Pain as bad as you can imagine.
Time Frame: 48 hours
Population: Because the Sponsor terminated the study, the planned sample size was not reached in any treatment group, therefore, only a brief summary of an exploratory analysis of the primary efficacy variable (SPID48) is presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tapentadol IR Fixed Dose 50 mg | Tapentadol IR Fixed Dose 75 mg | Tapentadol IR Fixed Dose 100 mg | Oxycodone HCL IR Fixed Dose 10 mg | Placebo Fixed Dose
Number analyzed (Participants) | 35 | 31 | 30 | 36 | 24
score on a scale | 73.9 (123.89) | 54.4 (128.22) | 49.3 (136.92) | 57.6 (125.73) | -18.6 (130.74)
Statistical Analysis 1: Comparison: Tapentadol IR Fixed Dose 50 mg vs Placebo Fixed Dose; The study was terminated and did not reach the planned sample size; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference of SPID48 = 91.4, 95% CI [49.77 to 133.07]
Statistical Analysis 2: Comparison: Tapentadol IR Fixed Dose 75 mg vs Placebo Fixed Dose; The study was terminated and did not reach the planned sample size; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference of SPID48 = 81.5, 95% CI [38.66 to 124.29]
Statistical Analysis 3: Comparison: Tapentadol IR Fixed Dose 100 mg vs Placebo Fixed Dose; The study was terminated and did not reach the planned sample size; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference of SPID48 = 81.5, 95% CI [39.21 to 123.80]
Statistical Analysis 4: Comparison: Oxycodone HCL IR Fixed Dose 10 mg vs Placebo Fixed Dose; The study was terminated and did not reach the planned sample size; Test type: Superiority or Other; p < 0.001, ANCOVA; LS mean difference of SPID48 = 82.4, 95% CI [38.96 to 125.88]

2. Secondary Outcome: Time to First Rescue Pain Medication.
Time Frame: 3 days
Population: Due to termination of trial, results were not analyzed.
Arm/Group | Tapentadol IR Fixed Dose 50 mg | Tapentadol IR Fixed Dose 75 mg | Tapentadol IR Fixed Dose 100 mg | Oxycodone HCL IR Fixed Dose 10 mg | Placebo Fixed Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: The SPID at 12, 24, and 72 Hours Relative to First Dose.
Description: The SPID score incorporates the cumulative analgesic effects of tapentadol IR on pain intensity over an extended period (12 to 72 hours) allowing for an evaluation of multiple doses of drug, even when dosing frequency may vary. Scoring is derived from the Numerical Rating Scale (NRS) from 0 = No pain to 11 = Pain as bad as you can imagine.
Time Frame: 3 days
Population: Due to termination of trial, results were not analyzed.
Arm/Group | Tapentadol IR Fixed Dose 50 mg | Tapentadol IR Fixed Dose 75 mg | Tapentadol IR Fixed Dose 100 mg | Oxycodone HCL IR Fixed Dose 10 mg | Placebo Fixed Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated informed consent was obtained throughout the follow-up phase of the study. Serious adverse events were collected for 30 days after the last dose of study drug.
Arm/Group | Tapentadol IR Fixed Dose 50 mg | Tapentadol IR Fixed Dose 75 mg | Tapentadol IR Fixed Dose 100 mg | Oxycodone HCL IR Fixed Dose 10 mg | Placebo Fixed Dose
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/71 | 3/75 | 1/67 | 0/75
Other Adverse Events (participants affected / at risk) | 52/77 | 38/71 | 53/75 | 43/67 | 44/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol IR Fixed Dose 50 mg (N=77) | Tapentadol IR Fixed Dose 75 mg (N=71) | Tapentadol IR Fixed Dose 100 mg (N=75) | Oxycodone HCL IR Fixed Dose 10 mg (N=67) | Placebo Fixed Dose (N=75)
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol IR Fixed Dose 50 mg (N=77) | Tapentadol IR Fixed Dose 75 mg (N=71) | Tapentadol IR Fixed Dose 100 mg (N=75) | Oxycodone HCL IR Fixed Dose 10 mg (N=67) | Placebo Fixed Dose (N=75)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 8 | 11 | 7
Body Temperature Increased (Investigations) | 8 | 7 | 4 | 5 | 7
Confusional State (Psychiatric disorders) | 6 | 4 | 11 | 1 | 0
Constipation (Gastrointestinal disorders) | 11 | 6 | 10 | 12 | 7
Dizziness (Nervous system disorders) | 7 | 8 | 16 | 14 | 4
Dry Mouth (Gastrointestinal disorders) | 1 | 7 | 3 | 3 | 0
Hallucination, Visual (Psychiatric disorders) | 2 | 5 | 8 | 2 | 2
Headache (Nervous system disorders) | 5 | 5 | 2 | 9 | 13
Hypotension (Vascular disorders) | 4 | 1 | 5 | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 3 | 1 | 3 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 19 | 5 | 12 | 12 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 4 | 0
Pyrexia (General disorders) | 15 | 8 | 13 | 14 | 7
Somnolence (Nervous system disorders) | 11 | 10 | 17 | 6 | 1
Vomiting (Gastrointestinal disorders) | 5 | 6 | 4 | 10 | 12

LIMITATIONS AND CAVEATS:
Sponsor terminated study, sample size not reached. The protocol section describes 4 study arms defining the treatment groups in the study design. The participant flow module describes the 5 treatment groups analyzed for the primary endpoint

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A provision provides for 60 day prior review by sponsor extendable by 60 days to file a patent application and prior written consent of sponsor for disclosure of confidential information, if any.